CLINICAL TRIAL: NCT00180908
Title: SFOP-OS94: Multicentric Randomised Phase III Trial Comparing Efficacy of Preoperative High-Dose Methotrexate Plus Doxorubicin to Efficacy of High-Dose Methotrexate Plus Etoposide and Ifosfamide, in Children and Adolescents Osteosarcoma
Brief Title: Comparison of High-Dose Methotrexate (HDM) Plus Doxorubicin to HDM Plus Etoposide-Ifosfamide in Osteosarcoma Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS94; CSET-94-300
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Osteosarcoma; Localised High Grade Osteosarcoma of the Limbs
Keywords: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — IMVP-16 protocol; Doxorubicin; Methotrexate

INTERVENTIONS:
Drug: Etoposide, Ifosfamide, Methotrexate
Drug: Doxorubicin, Methotrexate

SUMMARY:
The purpose of this study is to compare two preoperative chemotherapy regimens based on high-dose methotrexate courses given alternately either with doxorubicin or with etoposide-ifosfamide.

ELIGIBILITY:
Inclusion Criteria:

* non metastatic limb osteosarcoma,
* age less than 20 years,
* biopsy proven high-grade osteosarcoma,
* no previous treatment,
* no contraindication to chemotherapy
* no previous malignancy,
* Written informed consent.

Exclusion Criteria:

* juxta-cortical sarcoma and microcellular anaplastic sarcoma,
* previous anticancer treatment
* contraindication to chemotherapy
* previous malignancy,

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226
Dates: Start 1994-06

PRIMARY OUTCOMES:
Good histological response (5% or less viable cells) after preoperative chemotherapy

SECONDARY OUTCOMES:
Event-free survival,
Overall survival,
Toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Kalifa, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Le Deley MC, Guinebretiere JM, Gentet JC, Pacquement H, Pichon F, Marec-Berard P, Entz-Werle N, Schmitt C, Brugieres L, Vanel D, Dupouy N, Tabone MD, Kalifa C; Societe Francaise d'Oncologie Pediatrique (SFOP). SFOP OS94: a randomised trial comparing preoperative high-dose methotrexate plus doxorubicin to high-dose methotrexate plus etoposide and ifosfamide in osteosarcoma patients. Eur J Cancer. 2007 Mar;43(4):752-61. doi: 10.1016/j.ejca.2006.10.023. Epub 2007 Jan 30. PMID 17267204